CLINICAL TRIAL: NCT02388152
Title: Interventional, Open-label, Multiple-immunization Extension Study on the Safety, Tolerability and Immunogenicity of Lu AF20513/Adjuvant in Patients With Alzheimer's Disease
Brief Title: Study to Evaluate the Safety and Tolerability of a New Drug Named Lu AF20513 in Patients With Mild Alzheimer's Disease
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: New data: The study was terminated based on new efficacy data from another study
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16026A; 2014-001797-34 (EudraCT Number)
Record Dates: First submitted 2015-03-03; First posted 2015-03-13 (Estimated); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Lu AF20513, low dose (Cohort 1) (Experimental): 10 Patients with mild Alzheimer's.
  Interventions: Drug: Lu AF20513, low dose
- Lu AF20513, medium dose (Cohort 2) (Experimental): 10 Patients with mild Alzheimer's.
  Interventions: Drug: Lu AF20513, medium dose
- Lu AF20513, high dose (Cohort 3) (Experimental): 15 Patients with mild Alzheimer's.
  Interventions: Drug: Lu AF20513, high dose
- Lu AF20513, double high dose (Cohort 4) (Experimental): 15 Patients with mild Alzheimer's.
  Interventions: Drug: Lu AF20513, double high dose

INTERVENTIONS:
Drug: Lu AF20513, low dose
  Arms: Lu AF20513, low dose (Cohort 1)
Drug: Lu AF20513, medium dose
  Arms: Lu AF20513, medium dose (Cohort 2)
Drug: Lu AF20513, high dose
  Arms: Lu AF20513, high dose (Cohort 3)
Drug: Lu AF20513, double high dose
  Arms: Lu AF20513, double high dose (Cohort 4)

SUMMARY:
The purpose of this study is to determine if multiple immunizations with Lu AF20513 is tolerable and safe in patients with mild Alzheimer's disease.

ELIGIBILITY:
Main Inclusion Criteria:

* The patient has a diagnosis of probable Alzheimer's Disease (AD) consistent with the National Institute of Neurological and Communicative Disorders and Stroke and the Alzheimer's Disease and Related Disorders Association (NINCDS-ADRDA) criteria
* The patient has a pattern of antibodies in cerebrospinal fluid (CSF) consistent with an amyloid plaque load
* The patient is a man or a woman, and between ≥60 and ≤85 years of age
* The patient has an MRI (performed within 3 months before screening) with results consistent with the diagnosis of probable AD
* The patient has a mild severity of dementia
* The patient has a knowledgeable and reliable caregiver who will be available and able to: accompany the patient to all clinical visits, monitor IRE after each immunization, and participate with the patient at all phone visits during the study AD
* Patients must have completed Part A before being eligible for continued immunisations in Part B

Main Exclusion Criteria:

* The patient has evidence of mixed etiology of dementia (i.e. absence of other neurodegenerative, neuroinflammatory or cerebrovascular disease, or another neurological, mental or systemic disease or condition likely contributing to cognitive decline)
* The patient has clinical and radiological findings that fulfil the standards of the National Institute of Neurological Disorders and Stroke and Association Internationale pour la Recherché et l'Enseignement en Neurosciences (NINDS-AIREN) criteria for vascular dementia
* The patient has a Diagnostic and Statistical Manual of Mental Disorders, 4th edition, Text Revision (DSM-5-TR) Axis I disorder other than AD; including amnestic disorders, delirium, schizophrenia or schizoaffective disorder, bipolar disorder, current major depressive episode, psychosis, panic, post-traumatic stress disorder and/or cognitive disorder not otherwise specified, (note: patients may be included if treated with a stable dose of antidepressants for at least 2 months and not fulfilling DSM-5-TR criteria for depression at Screening)
* The patient's eligibility MRI scan (1.5T) shows findings that correspond to more than 4 brain micro haemorrhages
* The patient has extensive white matter lesions as shown on the screening MRI scan (1.5T)

Other protocol-defined inclusion and exclusion criteria do apply

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-03; Primary Completion 2019-07-04 (Actual); Study Completion 2019-07-04 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability assessed by composite outcome measure consisting of absolute values and changes from baseline in: adverse events, clinical safety laboratory tests, vital signs | Baseline to week 96
  ECGs, physical and neurological examination, suicidality assessment, Immunisation-Related Events (IRE) (selected from Brighton Collaboration guidelines) and magnetic resonance imaging (MRI) safety scans
Antibody titre | Baseline to week 96

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (5):
- AT001, Vienna, Austria
- FI001, Turku, Finland
- Sweden (3):
  - SE002, Malmo
  - SE003, Mölndal
  - SE001, Stockholm